CLINICAL TRIAL: NCT01233999
Title: Botulinum Toxin in the Treatment of Raynaud's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suephy Chen, MD, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00015510
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Raynaud's Syndrome
Keywords: Scleroderma; Raynaud's Syndrome
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botox (Placebo Comparator): single-drug dosage comparison cross-over study
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — Botulinum toxin A will be injected into participants hand total 40units

SUMMARY:
The investigators are studying a medical condition known as Raynaud's Phenomenon (RP). RP is a painful condition in which cold surroundings or stressful events trigger pain, a cold sensation, and in severe cases, sores and ulcers on one's fingers. The investigators think that RP results from problems with some of the components of the blood vessels, surrounding nerves, and some of the circulating messengers in the bloodstream. Although there are many different medicines that are currently used to treat RP, the investigators have not yet found a cure for severe cases of this condition. Furthermore, the investigators have found few medicines that show consistent healing of the ulcers that may be associated with RP. Some of the treatments include medicines that are used to treat high blood pressure known as calcium channel blockers. Medications that thin the blood (anticoagulants) such as aspirin have also been used to treat RP.

In this study, the investigators will investigate a new treatment for RP known as Botulinum toxin A. Botulinum toxin is a chemical that is temporarily toxic to nerves, but has been approved by the government for the treatment of several other conditions including but not limited to: excessive sweating, neck pain associated with a condition known as cervical dystonia, uncontrollable forcible closure of the eyelids known as blepharospasm, and a condition known as strabismus in which the eyes are not in alignment with one another.

This study will aim to greatly improve the quality of life and pain associated with RP. Previous studies also support the chance that Botulinum toxin will help to heal some of the ulcers associated with RP. Although there is no current standard of care, many of the patients in the study will have already failed or are unable to tolerate commonly used treatments such as lifestyle modifications, calcium channel blockers, nitroglycerin, and anticoagulants. If the patient chooses to participate in the study, he/she will be randomly assigned to receive an injection with Botulinum toxin in either the left or right hand. The other hand will be injected with saline solution. Neither the patient nor the physician or research personnel seen in follow-up will know which hand is injected with Botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:Adult (>18 years) patients with severe RP of any etiology will be invited to participate. Inclusion criteria include a) history of digital infarcts or ulcerations, b) unresponsive to standard therapies, or c) impending potential for digital amputation. Patients on other standard therapies such as antiplatelet agents, vasodilators, and calcium channel blockers will be included. -

Exclusion Criteria:Pregnancy, mild disease, patients with myasthenia gravis, botulinum toxin allergy, and phobia of needles are exclusion criteria. Women of childbearing age will need to demonstrate a negative urine pregnancy test. Myasthenia gravis is excluded because underlying generalized weakness can be exacerbated, and local weakness at injection sites can occur more than otherwise expected.

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suephy C Chen, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 subjects recruited from Emory Dept of Dermatology
Pre-assignment Details: all subjects were assigned to group
Groups:
- Botox: Participants will be randomly assigned to receive 1 injection with Botulinum toxin A, 40 units in either the left or right hand.
Period: Overall Study
Arm/Group | Botox
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Botox
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Digital Temperature Difference From Baseline
Description: Each digit temperature was measured and recorded at baseline, and then measured and re-recorded after 3 minute intervals following a 20 second 4 degree Celsius ice bath immersion.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Celsius
Arm/Group | Botox
Number analyzed (Participants) | 9
Celsius | 1.30 [0.23 to 2.36]

ADVERSE EVENTS:
Description: A total of 10 participants signed the informed consent, 8 participants completed the trial, 1 participant received study drug and became lost to follow-up and one participant withdrew consent prior to receiving an injection.
Arm/Group | Botox
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Pilot study with limited numbers to analyze

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No